CLINICAL TRIAL: NCT02151851
Title: A Phase 3, Multi-center, Double-blind, Placebo-controlled, Parallel Group, Randomized 24-week Study to Evaluate the Safety and Efficacy of Certolizumab Pegol (CZP) as Additional Medication to Methotrexate in Chinese Subjects With Active Rheumatoid Arthritis Who Have an Incomplete Response to Methotrexate
Brief Title: A Study of Certolizumab Pegol as Additional Therapy in Chinese Patients With Active Rheumatoid Arthritis
Acronym: RAPID-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA, Belgium (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RA0044
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; TNFα antagonist; Certolizumab Pegol; Chinese patients
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Certolizumab Pegol + Methotrexate (Experimental): Subjects will receive loading doses of CZP 400 mg (200 mg / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then CZP 200 mg (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
  Interventions: Biological: Certolizumab Pegol; Drug: Methotrexate
- Placebo + Methotrexate (Placebo Comparator): Subjects will receive Placebo (1mL / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then Placebo (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
  Interventions: Drug: Methotrexate; Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active substance: Certolizumab Pegol
  * Pharmaceutical Form: Prefilled syringes
  * Concentration: 200 mg/ml
  * Route of administration: Subcutaneous injection
  Other Names: Cimzia
  Arms: Certolizumab Pegol + Methotrexate
Drug: Methotrexate — * Active substance: Methotrexate
  * Pharmaceutical form: Tablet
  * Concentration: Maximum dose 10 mg per week
  * Route of administration: Oral
Other: Placebo — * Active substance: Placebo
  * Pharmaceutical form: Prefilled syringes
  * Concentration: 0.9 % saline
  * Route of Administration: Subcutaneous injection
  Arms: Placebo + Methotrexate

SUMMARY:
This study will evaluate the safety & efficacy of Certolizumab Pegol (CZP) as additional medication to Methotrexate (MTX) in Chinese subjects with Rheumatoid Arthritis. 400 patients will be randomized to receive either CZP + MTX or placebo + MTX. Anticipated time in the study is about 32 weeks.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, double-blind, placebo-controlled, parallel group, randomized, 24-week study to evaluate the safety and efficacy of Certolizumab Pegol (CZP) as additional medication to Methotrexate (MTX) in Chinese subjects with active Rheumatoid Arthritis (RA) who have an incomplete response to Methotrexate. This study is designed to determine whether CZP 400 mg at Weeks 0, 2, and 4 followed by CZP 200 mg every 2 weeks (Q2W) in combination with MTX demonstrates superiority, in terms of greater improvement in relief of the signs and symptoms of RA, compared with MTX alone. Approximately 535 subjects will be screened to randomize 400 subjects into this study, at approximately 25 centers in the People's Republic of China. There will be 2 treatment groups, with 300 subjects in the CZP+MTX group and 100 subjects in the PBO+MTX group. For each subject, the study duration will last a maximum of approximately 38 weeks. Subjects who complete study RA0044 and subjects who fail to achieve an American College of Rheumatology 20 % Response Criteria (ACR20) response at Week 12 that is confirmed at Week 14 and thus are withdrawn from this study at Week 16, are permitted to receive treatment with CZP in the open-label extension study, RA0078. The secondary objectives are to assess the dose regimen of CZP in combination with MTX compared with MTX alone in the safety and tolerability, ability to improve physical function, and health outcomes measures in Chinese subjects with active RA; also to characterize the pharmacokinetic (PK) profile and immunogenicity of CZP in combination with MTX.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form (ICF) is signed and dated by the subject or by the legal representative
* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete questionnaires), visit schedule, and medication intake according to the judgment of the Investigator
* Subject is male or female, and at least 18 years of age at the Screening Visit
* Subjects must have a diagnosis of adult onset Rheumatoid Arthritis RA of at least 6 months duration as defined by the 1987 American College of Rheumatology (ACR) classification criteria (Arnett et al, 1988).
* Subjects must have active RA disease as defined by:

  * ≥6 tender joints at Screening and Baseline
  * ≥6 swollen joints at Screening and Baseline
  * Fulfilling 1 of the following 2 criteria during the Screening Period:
  * European League Against Rheumatism (ESR) (Westergren) ≥30 mm/hour, or
  * C-reactive protein (CRP) >15 mg/L
* Subjects must have a normal chest x ray within 3 months prior to the Baseline Visit
* Female subjects with childbearing potential should have a negative pregnancy test at Screening and at Baseline and should have a medically accepted method of contraception used during the entire duration of the study and for 10 weeks after the last dose of Certolizumab Pegol (CZP).
* Male subjects must agree to ensure they use adequate contraception during the study and for at least 10 weeks after the subject receives their last dose of study medication
* Subjects must have received treatment with Methotrexate (MTX) (with or without folic acid) for at least 3 months prior to the Baseline Visit. The dose and route of administration of MTX must have been stable for at least 2 months prior to the Baseline Visit. The minimum stable dose of MTX allowed is 10 mg weekly

Exclusion Criteria:

Rheumatoid Arthritis disease-related exclusions:

* Subjects have a diagnosis of any other inflammatory arthritis (eg, psoriatic arthritis or ankylosing spondylitis)
* Subjects have a secondary, noninflammatory type of arthritis (eg, Osteoarthritis or Fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of study medication on the subject's primary diagnosis of Rheumatoid Arthritis (RA)
* Subjects have a history of an infected joint prosthesis at any time with that prosthesis still in situ
* Subjects have >3 arthroplasties due to RA and/or Steinbrocker IV functional capacity

Concomitant medication exclusions:

* Subjects must be free of prohibited medication, Analgesics (including Paracetamol and Acetominophen), NSAIDs /COX-2 Inhibitors, Oral corticosteroids, DMARDs, etc. as detailed in protocol Previous clinical studies and previous biological therapy exclusions
* Subjects have previously participated in this study or subject has previously been assigned to treatment in a study of the medication under investigation in this study
* Subjects have participated in another study of an investigational medicinal product (or a medical device) within the previous 3 months or are currently participating in another study of an investigational medicinal product (or a medical device)
* Subjects have received any experimental nonbiological therapy, within or outside a clinical study in the 3 months or within 5 half lives (whichever is longer) prior to Baseline Visit
* Subjects have received any biological therapy for RA within 3 months or within 5 half lives (whichever is longer) prior to Baseline Visit, except for Etanercept and Anakinra where only a 1 month washout prior to the Baseline Visit is necessary
* Subjects have received Rituximab or Tocilizumab
* Subjects have received Yunke (technetium-99 conjugated with methylene diphosphonate) other than for diagnostic purpose within 5 years prior to Baseline
* Subjects have received previous treatment with a biological therapy for RA that resulted in a severe hypersensitivity reaction or an anaphylactic reaction
* Subjects who failed to respond to previous treatment with a Tumor Necrosis Factor (TNF) blocking drug are excluded. Subjects who initially responded to a maximum of 2 TNF blocking agents but who later discontinued the agent(s) due to loss of efficacy or other reasons may be included

Medical history exclusions:

* Female subjects who are breast feeding, pregnant, or plan to become pregnant during the study or for 3 months following last dose of study medication
* Subjects with a history of chronic infection, recent serious or life threatening infection (within 6 months, including herpes zoster), or a current sign or symptom that may indicate an infection (eg, fever, cough)
* Subjects with a history or active systemic/respiratory infection due to fungal, parasitic, or mycotic pathogens including but not limited to histoplasmosis, coccidiosis, paracoccidiosis, pneumocystis, blastomyces, aspergillus, and nontuberculous mycobacteria (NTMB)
* Radiographic evidence suggestive of any of these infections is sufficient grounds for exclusion
* Subjects with known Tuberculosis (TB) infection, at high risk of acquiring TB infection, or Latent Tuberculosis (LTB) infection are excluded
* Subjects at a high risk of infection (eg, leg ulcers, indwelling urinary catheter, persistent or recurrent chest infections, and subjects that are permanently bedridden or wheelchair bound)
* Subjects with a positive Hepatitis B surface antigen (HBsAg) test and/or Hepatitis C virus antibody (anti HCV) test result
* Subjects with positive human immunodeficiency virus (HIV) test
* Subjects receiving any live (includes attenuated) vaccination within 56 days prior to Baseline (eg, injectable influenza and pneumococcal vaccines are allowed, but nasal influenza vaccine is not)
* Subjects with a history of a lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoproliferative disease at any time
* Subjects with an active malignancy of any type or a history of malignancy (other than carcinoma of the cervix or basal cell carcinoma successfully treated more than 5 years prior to Screening)
* Subjects with a history of blood dyscrasias, eg, leukemia or hemophilia where the blood constituents are abnormal or are present in abnormal quantity
* Subjects with class III or IV congestive heart failure New York Heart Association (NYHA) 1994
* Subjects with a history of, or suspected, demyelinating disease of the central nervous system (eg, multiple sclerosis or optic neuritis)
* Subjects with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, GI, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the subject's participation in the study. Abnormal laboratory parameters as detailed in protocol that require exclusion of a subject
* Subjects with a history of an adverse reaction to Polyethylene Glycol (PEG) or a protein based medicinal product or known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB Pharma
Locations (30):
- China (30):
  - 037, Baotou
  - 001, Beijing
  - 002, Beijing
  - 013, Beijing
  - 021, Beijing
  - 025, Beijing
  - 033, Beijing
  - 014, Bengbu
  - 011, Changchun
  - 034, Changchun
  - 017, Changsha
  - 019, Changsha
  - 007, Chengdu
  - 012, Chengdu
  - 004, Guangzhou
  - 015, Hangzhou
  - 008, Harbin
  - 005, Hefei
  - 022, Jinan
  - 031, Kunming
  - 028, Nanjing
  - 009, Shanghai
  - 018, Shanghai
  - 020, Shanghai
  - 030, Shanghai
  - 038, Shijiazhuang
  - 010, Tianjin
  - 006, Wuhan
  - 016, Xi'an
  - 035, Xi'an

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in July 2014 and concluded in June 2016.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Period: Overall Study
Arm/Group | Placebo + Methotrexate | Certolizumab Pegol + Methotrexate
Started | 114 | 316
Included in the Safety Set | 113 | 316
Completed | 38 | 186
Not Completed | 76 | 130
Not completed — Lack of Efficacy | 67 | 94
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Medical impairment | 1 | 0
Not completed — Low compliance to study visits | 0 | 1
Not completed — Subject entered into study in error | 0 | 1
Not completed — Adverse Event | 6 | 28

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all subjects who received at least 1 dose of study medication.
Arm/Group | Placebo + Methotrexate | Certolizumab Pegol + Methotrexate | Total Title
Number analyzed (Participants) | 113 | 316 | 429
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 298 | 405
  >=65 years | 6 | 18 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.1) | 48.2 (11.8) | 47.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 268 | 363
  Male | 18 | 48 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 24
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 24 in the number of tender joints, in the number of swollen joints, and a 20 % or greater improvement in at least 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least 1 dose of study medication administration and provided any efficacy data after the first administration.
  NRI = non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Placebo + Methotrexate (FAS): Subjects will receive Placebo (1mL / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then Placebo (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
- Certolizumab Pegol + Methotrexate (FAS): Subjects will receive loading doses of CZP 400 mg (200 mg / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then CZP 200 mg (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
Arm/Group | Placebo + Methotrexate (FAS) | Certolizumab Pegol + Methotrexate (FAS)
Number analyzed (Participants) | 113 | 312
percentage of participants | 23.9 | 54.8
Statistical Analysis 1: Comparison: Placebo + Methotrexate (FAS) vs Certolizumab Pegol + Methotrexate (FAS); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Difference of CZP + MTX versus Placebo + MTX (and corresponding p-value) was estimated from a logistic regression model with factors for treatment and region; Odds Ratio (OR) = 3.899, 95% CI 2-sided [2.382 to 6.382]

2. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 24
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 24 in the number of tender joints, in the number of swollen joints, and a 50 % or greater improvement in at least 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Methotrexate (FAS) | Certolizumab Pegol + Methotrexate (FAS)
Number analyzed (Participants) | 113 | 312
percentage of participants | 7.1 | 36.5
Statistical Analysis 1: Comparison: Placebo + Methotrexate (FAS) vs Certolizumab Pegol + Methotrexate (FAS); Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.641, 95% CI 2-sided [3.570 to 16.352]

3. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 24
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 24 in the number of tender joints, in the number of swollen joints, and a 70 % or greater improvement in at least 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Methotrexate (FAS) | Certolizumab Pegol + Methotrexate (FAS)
Number analyzed (Participants) | 113 | 312
percentage of participants | 2.7 | 16.7
Statistical Analysis 1: Comparison: Placebo + Methotrexate (FAS) vs Certolizumab Pegol + Methotrexate (FAS); Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.248, 95% CI 2-sided [2.209 to 23.786]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 24
Description: The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions. Each domain consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3. A total score is computed from the item scores using the scoring rules provided by the index's author. HAQ-DI scores range from 0 to 3. Lower scores indicate less disability. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least 1 dose of study medication administration and provided any efficacy data after the first administration.
  LOCF = last observation carried forward. Only subjects with available HAQ-DI scores at week 24 were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Methotrexate (FAS) | Certolizumab Pegol + Methotrexate (FAS)
Number analyzed (Participants) | 110 | 306
units on a scale | -0.185 (0.463) | -0.530 (0.589)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) up to Week 25.
Description: Adverse Events refer to the Safety Set which consists of all subjects who received at least 1 dose of study medication.
Groups:
- Placebo + Methotrexate (SS): Subjects will receive Placebo (1mL / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then Placebo (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
- Certolizumab Pegol + Methotrexate (SS): Subjects will receive loading doses of CZP 400 mg (200 mg / prefilled syringe [PFS], ie, 2 injections) at Baseline, and Weeks 2 and 4; then CZP 200 mg (1 injection) Q2W until Week 22.
  All subjects will continue their treatment on Methotrexate (MTX), with or without folic acid, at the same dose and route of administration as at entry (unless there is a need to reduce the dose for reasons of toxicity, minimum dose permitted 10 mg per week).
Arm/Group | Placebo + Methotrexate (SS) | Certolizumab Pegol + Methotrexate (SS)
Serious Adverse Events (participants affected / at risk) | 3/113 | 20/316
Other Adverse Events (participants affected / at risk) | 48/113 | 130/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Methotrexate (SS) (N=113) | Certolizumab Pegol + Methotrexate (SS) (N=316)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Pericarditis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Methotrexate (SS) (N=113) | Certolizumab Pegol + Methotrexate (SS) (N=316)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 17 (19)
Upper respiratory tract infection (Infections and infestations) | 15 (21) | 50 (60)
Latent tuberculosis (Infections and infestations) | 7 (7) | 24 (24)
Urinary tract infection (Infections and infestations) | 7 (11) | 13 (18)
Liver function test abnormal (Investigations) | 4 (6) | 22 (24)
Alanine aminotransferase increased (Investigations) | 8 (9) | 19 (26)
White blood cell count decreased (Investigations) | 1 (1) | 18 (24)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 16 (18)
Neutrophil count increased (Investigations) | 8 (12) | 6 (6)
Lymphocyte count decreased (Investigations) | 8 (11) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days